CLINICAL TRIAL: NCT06021821
Title: A Randomized-Controlled Trial to Investigate the Effect of a Novel Music Therapy Application to Reduce Anxiety and Stress
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: SoundMind (Industry)
Collaborators: Citruslabs (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 20288
Record Dates: First submitted 2023-08-27; First posted 2023-09-01 (Actual); Last update posted 2023-09-01 (Actual); Status verified 2023-08

CONDITIONS: Anxiety; Depression; Stress
MeSH Terms: conditions — Anxiety Disorders; Depression

STUDY DESIGN:
Intervention Model Description: Three-group study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Intervention Group (Experimental): Participants will listen to the SoundMind app for 20 minutes per day, ideally during a moment of stress.
  Interventions: Other: SoundMind App
- Spotify Group (Active Comparator): Participants will listen to a specified Spotify playlist for 20 minutes per day, ideally during a moment of stress.
  Interventions: Other: Spotify Playlist
- Control Group (No Intervention): This group will have no tasks prescribed.

INTERVENTIONS:
Other: SoundMind App — he SoundMind application uses binaural beats to encourage relaxation, focus, and alertness.
  Arms: Intervention Group
Other: Spotify Playlist — Participants will listen to a "calm vibes" playlist by Spotify.
  Arms: Spotify Group

SUMMARY:
This virtual, open-label, three-group, randomized-controlled trial will last six weeks. Participants will be allocated into three groups; the Intervention Group, Spotify Group, and Control Group. All participants will complete a baseline questionnaire before completing their designated regime daily for six weeks. In addition, participants will complete study-specific surveys and validated questionnaires at the end of each week (Week 1, 2, 3, 4, 5 & 6). The study will include 75 [participants in total, 25 per group, who all have self-reported concerns around anxiety, stress, or depression.

Questionnaires will be used to monitor sleep, cognitive ability, and changes in symptoms of anxiety, depression, and stress. Both study-specific questionnaires and validated questionnaires will be utilized, including the Generalized Anxiety Disorder Assessment (GAD-7), the 9-question Patient Health Questionnaire (PHQ-9), Perceived Stress Scale (PSS), and The World Health Organisation- Five Well-Being Index (WHO-5). Likert scale responses will be examined from baseline to each check-in. Participant responses on product feedback will be presented as % scores.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* Between 18-28 years of age
* Self-reported concerns around anxiety, stress, or depression
* Generally healthy - don't live with any uncontrolled chronic disease
* Must have headphones

Exclusion Criteria:

* Any pre-existing chronic conditions that would prevent participants from adhering to the protocol, including oncological and psychiatric disorders
* Women who are pregnant, breastfeeding or attempting to become pregnant
* Unwilling to follow the study protocol
* Testing any other product for any other research studies at the same time
* History of epilepsy or seizures

Ages: 18 Years to 28 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 75 (Actual)
Dates: Start 2023-05-29 (Actual); Primary Completion 2023-07-26 (Actual); Study Completion 2023-07-26 (Actual)

PRIMARY OUTCOMES:
Change in scores on the Generalized Anxiety Disorder 7-item scale (GAD-7). [Baseline to Week 6] | 6 weeks
  The GAD-7 is a self-report questionnaire used to assess the severity of generalized anxiety disorder. It consists of seven questions that ask about the frequency and intensity of common symptoms of anxiety over the past two weeks. Each question is scored on a scale from 0 to 3, with the total scores ranging from 0 to 21. The scoring is typically interpreted as follows:
  0-4: Minimal anxiety 5-9: Mild anxiety 10-14: Moderate anxiety 15-21: Severe anxiety
Change in scores on the Patient Health Questionnaire-9 (PHQ-9). [Baseline to Week 6] | 6 weeks
  The PHQ-9 is a self-report questionnaire used to assess the severity of depression symptoms. Each question is scored on a scale from 0 to 3, with the total scores ranging from 0 to 27. The scoring is typically interpreted as follows:
  0-4: Minimal depression 5-9: Mild depression 10-14: Moderate depression 15-19: Moderately severe depression 20-27: Severe depression
Change in scores on the Perceived Stress Scale (PSS). [Baseline to Week 6] | 6 weeks
  The PSS is a widely used self-report questionnaire designed to measure an individual's perception of stress in their life. Higher scores indicate higher perceived stress.
Change in scores on the World Health Organization Well-Being Index (WHO-5). [Baseline to Week 6] | 6 weeks
  The WHO-5, or World Health Organization Well-Being Index, is a self-reported questionnaire used to measure psychological well-being and mood. Respondents are asked to rate statements on a scale from 0 to 5, where 0 indicates "at no time" and 5 indicates "all of the time." The scores are summed, resulting in a total score that can range from 0 to 25. A total score of 0-13 suggests poor well-being and a higher risk of depression.
  A total score of 14-17 indicates moderate well-being. A total score of 18-25 suggests good well-being.

SECONDARY OUTCOMES:
Changes in participant-perceived sleep quality. [Baseline to Week 6] | 6 weeks
  Survey-based assessment of participants' perception of their sleep quality.

CONTACTS AND LOCATIONS:
Locations (1):
- Citruslabs, Santa Monica, California, United States

IPD SHARING:
Plan to Share IPD: Undecided